CLINICAL TRIAL: NCT05915325
Title: Physical Training for Elderly Cancer Patients With Cachexia (TEECH-01): a Prospective Clinical Trial
Brief Title: Physical Training for Elderly Cancer Patients With Cachexia
Acronym: TEECH-01
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Collaborators: National Cheng Kung University (Other)
Responsible Party: Principal Investigator, Chih Chieh, Yen, Principal investigator, National Cheng-Kung University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TEECH-01
Record Dates: First submitted 2023-05-20; First posted 2023-06-23 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Geriatric Assessment; Cancer; Cancer Cachexia
Keywords: Geriatric cancer; Cancer cachexia; Physical training; Severity
MeSH Terms: conditions — Neoplasms | interventions — Physical Conditioning, Human

STUDY DESIGN:
Intervention Model Description: Single-arm intervention trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physical training (Experimental): Supervised patient-tailored intensity-modulated physical training
  Interventions: Procedure: Physical training

INTERVENTIONS:
Procedure: Physical training — 1. Supervised Physical Training in SeniorGym for 12 weeks: 1) Aerobic exercise: Patient-tailored intensity-modulated ergometer training for the limbs; 2) Resistance exercise: Patient-tailored resistance exercise by Theraband for the limbs
  2. Nutrition intervention for 24 weeks: Dietitian consultation, education and intervention for 24 weeks

SUMMARY:
The goal of the clinical trial is to evaluate the feasibility and efficacy of physical training for elderly cancer patients at risk of cancer cachexia. The main questions it aims to answer are:

* Whether a physical training program is feasible in elderly cancer patients with cachexia?
* What is the efficacy of a physical training program in reducing the severity of cancer cachexia in elderly cancer patients?

Participants will receive a 12-week supervised patient-tailored intensity-modulated physical training and being assessed for the severity of cancer cachexia before and after the training.

DETAILED DESCRIPTION:
The trial is to investigate the feasibility and efficacy of an artificial intelligence-based patient-tailored intensity-modulated physical training for cancer patients aged over 65 at risk of cancer cachexia. The primary endpoint is simplified cancer CAchexia SCOre (MiniCASCO) reduction. Secondary endpoints include geriatric assessment, physical activity and sarcopenia. This is an open-label, single-arm, single-center phase II investigator-initiated trial. The investigators assume a reduction of MiniCASCO by 10% after trial intervention. Under a statistical power of 80% and a probability of type I error at 0.1 (two-tailed), a minimal of 49 participants will be enrolled. All participants will receive a 12-week supervised physical training and nutritional intervention. Efficacy assessments will be conducted at baseline (week 0), post-intervention (week 12) and follow-up period (week 24). The investigators anticipate that the optimal patient-tailored training program is feasible and improves the symptoms and severity of elderly cancer cachexia. The results may shed light on the debilitating and burdensome condition and provide information on future clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged equivalent to or over 65 years with an existing cancer requiring antineoplastic treatments at trial enrollment, as defined by presence of a catastrophic disease certificate for malignancy in National Health Insurance (NHI)-Taiwan.
2. Subjects receive at least one systemic antineoplastic treatment within 12 weeks since trial enrollment, which includes chemotherapy, immunotherapy, hormonal, targeted and cellular therapy of whichever initial therapeutic intent (curative, palliative or salvage).
3. Subjects fulfill either cancer cachexia or pre-cachexia. (3.1) Cancer cachexia: A maximal weight loss of at least 5% from the baseline within 6 months in those whose BMI equivalent to or over 20 kg/m2 or at least 2% in those whose BMI less than 20 kg/m2; (3.2) Pre-cachexia: A maximal weight loss of 1% to 5% from the baseline within 6 months in patients whose BMI equivalent to or over 20 kg/m2 or 1% to 2% in those whose BMI less than 20 kg/m2 plus any of the following: an elevated serum C-reactive protein above upper normal limits (ULN), impaired fasting glucose or known diabetes mellitus, use of high-dose corticosteroid (over 10 mg prednisone equivalent daily), hypogonadism (disease-related or iatrogenic) or insufficient calorie intake of less than 20 kcal/kg/day
4. Subjects are in a clinical status with an expected life span exceeding 6 months and Eastern Cooperative Oncology Group (ECOG) 0 to 1 or Karnofsky Performance Scale (KPS) 80 to 100 at trial enrollment.
5. Subjects are physically and mentally capable and willing for conducting the planned physical training and agreed to comply the educational instructions and a wearable device during trial intervention.
6. Subjects are functionally and cognitively capable to be informed of the trial contents and objectives (including obtaining peripheral blood sampling for trial investigation), and agree to sign the written consent for enrollment.

Exclusion Criteria:

1. Subjects have tumor in situ or curatively treated malignant disease which requires no further antineoplastic treatments.
2. Subjects are anticipated to receive any surgery, radiotherapy or intervention that prevents or hinders a planned physical training within 28 weeks since trial enrollment.
3. Subjects experience a progressive body weight loss which fulfills the criteria for cancer cachexia or pre-cachexia but complicates with other confounding causes.
4. Subjects have cachexia caused by etiologies not limited to cancer.
5. Subject's malignant disease is considered unstable and thereby unfit for a planned physical training.
6. Subjects have an underlying medical illness causing severely impaired organ functions.
7. Subjects have an active infection requiring hospitalized treatment or intravenous anti-pathogen therapies.
8. Subjects who receive other experimental treatments or interventions for cancer cachexia.
9. Subjects are planning to conceive or already in pregnancy.
10. Subjects are currently participating in any other observational studies concerning cancer cachexia.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 23 (Actual)
Dates: Start 2023-07-05 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-01-05 (Estimated)

PRIMARY OUTCOMES:
Simplified cancer CAchexia SCOre (MiniCASCO) | Change from week 0 (trial enrollment) to week 12 (end of training)
  A simplified version for the scoring of the severity of cancer cachexia:
  A total score of 0 to 100 points are recorded and graded as minimal (0 to 14), mild (15 to 28), moderate (29 to 46) or severe cachexia (47 to 100)

SECONDARY OUTCOMES:
Integrated Care for Older People Guidelines score (ICOPE) | Change from week 0 (trial enrollment) to week 12 (end of training)
  Geriatric assessment:
  A total of 6 domains (cognitive, mobility, nutrition, visual, hearing and depressive symptoms) are included and be given a score of 1 on each if screened positive (a total score from 0 to 6). Of those who scored greater than 2 will be considered "impaired".
Physical Activity Performance Scale | Change from week 0 (trial enrollment) to week 12 (end of training)
  Hand grip strength, Gait speed, Body mass index, Sit-to-stand, Back stretch, Sit reach, Single leg stand, Up-and-go, 2-minute step, 6-minute walk test and Timed up-and-go:
  A total of 11 items will be recorded and calculated for the percentage difference, which is equivalent to the {[absolute change between week 12 (end of training) and week 0 (trial enrollment) testing result] / week 0 testing result } x 100 %. A mean percentage difference of the 11 items, ranging from 0 to 100%, will be calculated and of those with a greater mean percentage difference indicate a greater post intervention change.

OTHER OUTCOMES:
European Organisation for Research and Treatment of Cancer-Quality of Life Cancer C30 (EORTC-QLQ-C30) | Change from trial enrollment (week 0) to week 12 (end of training)
  Health-related quality of life:
  A total of 10 standardized questions from EORTC-QLQ C30 are asked to the participants. The answers are graded as none/not at all, a little/slightly, average/moderately, or a lot/considerably and each question is given 0, 0.25, 0.75 or 1.0 point, respectively. A sum-up score of 0 to 10 will be recorded and of those with a greater score indicate a poorer quality of life.
Mini Nutritional Assessment Short-Form (MNA-SF) | Change from trial enrollment (week 0) to week 12 (end of training)
  Nutrition:
  A total of six questions on food intake, weight loss, mobility, psychological stress/acute disease, the presence of dementia/depression, and body mass index will be graded. A total score, ranging from 0 to 14, will be recorded and of those with a score ≤ 11 indicate a nutritional deficit.

CONTACTS AND LOCATIONS:
Overall Officials: Chih Chieh Yen, MD, Principal Investigator — Department of Oncology, National Cheng Kung University Hospital
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No
The study protocol, statistical analysis plan and individual information are to be shared upon reasonable request to the study principal investigator.

REFERENCES:
- [Background] Poisson J, Martinez-Tapia C, Heitz D, Geiss R, Albrand G, Falandry C, Gisselbrecht M, Couderc AL, Boulahssass R, Liuu E, Boudou-Rouquette P, Chah Wakilian A, Gaxatte C, Pamoukdjian F, de Decker L, Antoine V, Cattenoz C, Solem-Laviec H, Guillem O, Medjenah H, Natella PA, Canoui-Poitrine F, Laurent M, Paillaud E. Prevalence and prognostic impact of cachexia among older patients with cancer: a nationwide cross-sectional survey (NutriAgeCancer). J Cachexia Sarcopenia Muscle. 2021 Dec;12(6):1477-1488. doi: 10.1002/jcsm.12776. Epub 2021 Sep 14. PMID 34519440
- [Background] Argiles JM, Betancourt A, Guardia-Olmos J, Pero-Cebollero M, Lopez-Soriano FJ, Madeddu C, Serpe R, Busquets S. Validation of the CAchexia SCOre (CASCO). Staging Cancer Patients: The Use of miniCASCO as a Simplified Tool. Front Physiol. 2017 Feb 17;8:92. doi: 10.3389/fphys.2017.00092. eCollection 2017. PMID 28261113
- [Background] Small SD, Bland KA, Rickard JN, Kirkham AA. Exercise-based Multimodal Programming: A Treatment Gap for Older Adults with Advanced Cancer. Oncologist. 2022 Feb 3;27(1):1-3. doi: 10.1093/oncolo/oyab009. PMID 35305110
- [Background] Arrieta H, Astrugue C, Regueme S, Durrieu J, Maillard A, Rieger A, Terrebonne E, Laurent C, Maget B, Servent V, Lavau-Denes S, Dauba J, Fonck M, Thiebaut R, Bourdel-Marchasson I. Effects of a physical activity programme to prevent physical performance decline in onco-geriatric patients: a randomized multicentre trial. J Cachexia Sarcopenia Muscle. 2019 Apr;10(2):287-297. doi: 10.1002/jcsm.12382. Epub 2019 Mar 4. PMID 30829460
- [Background] Mikkelsen MK, Lund CM, Vinther A, Tolver A, Johansen JS, Chen I, Ragle AM, Zerahn B, Engell-Noerregaard L, Larsen FO, Theile S, Nielsen DL, Jarden M. Effects of a 12-Week Multimodal Exercise Intervention Among Older Patients with Advanced Cancer: Results from a Randomized Controlled Trial. Oncologist. 2022 Feb 3;27(1):67-78. doi: 10.1002/onco.13970. PMID 34498352
- See also: Medical Device Innovation Center, National Cheng Kung University — https://mdic.ncku.edu.tw/
- See also: Geriatric Health Center, National Cheng Kung University Hospital — https://www.hosp.ncku.edu.tw/GH/about.html
- See also: Department of Computer Science and Information Engineering, National Cheng Kung University — https://www.csie.ncku.edu.tw/zh-hant/ncku_csie/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-01): https://cdn.clinicaltrials.gov/large-docs/25/NCT05915325/Prot_SAP_000.pdf